CLINICAL TRIAL: NCT00604448
Title: The Effect of Frequent Consumption of Pulses for Eight Weeks on Blood Lipids and on Glycemic and Satiety Hormones Response in Overweight and Obese Subjects
Brief Title: The Effect of Eating Pulses for 8 Weeks on Satiety and Metabolic Syndrome Risk Factors in Overweight Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pulse_Canada_481556; UfT fund#: 481556
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Overweight
Keywords: pulses; beans; obesity; overweight; metabolic syndrome
MeSH Terms: conditions — Obesity; Overweight; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulse group (Experimental): a group receiving a meal with pulses (5 cups/week) for 8 weeks
  Interventions: Other: Dietary advise; Other: Diet enriched with a meal containing pulses
- Energy-restricted group (Experimental): a group with a diet restriction of 500 kcal/day for 8 weeks
  Interventions: Other: Dietary advise; Other: Diet enriched with a meal containing pulses

INTERVENTIONS:
Other: Dietary advise — Subjects in energy-restricted group will follow dietician advise to keep a conventional energy restriction diet.
  Other Names: Energy-restricted group
Other: Diet enriched with a meal containing pulses — Subjects in pulse group will consume the commercially available pulses for 8 weeks
  Other Names: Pulse group

SUMMARY:
In 2004, almost 60% of adult Canadians were overweight or obese. This is a serious health concern due to the burden of common health risks associated with being overweight and obese, including increased blood sugar, blood lipids and blood pressure. Together these risks are known as metabolic syndrome. Obesity, the most common nutrition problem in Canada, can in many cases be treated through changes in our diet (what we eat and/or how much we eat). Pulses (beans, chickpeas, lentils and peas) when eaten on a regular basis may result in decreased health risks associated with being overweight and obese. The purpose of this study is to find out whether eating pulses (5 cups per week) results in improvements in metabolic syndrome risk factors. We also want to determine whether the consumption of pulses alters the levels of satiety hormones (hormones that make us feel hungry or full) in the blood. This study will have 50 participants.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effect of consuming 5 cups per week of commercially available pulses on body weight, satiety and metabolic syndrome risk factors in overweight/obese adults over 8 weeks with a conventional energy restriction diet.

The amount of pulses to be included in the study protocol is based on the USDA Dietary Guideline of 3 cups of pulses per week, but is somewhat high at 5 cups/week. Both groups will receive counseling from a registered dietitian. Pulses will be provided free of charge, delivered weekly to each participant and instructions will be given on their preparation. Subjects will be asked to complete a pulse log to record the date and time of day the pulses are consumed, as well as the type of pulse and other foods consumed during the pulse meal. Cooked pulses will be provided in canned or frozen forms. After completing the meal, subjects will be asked to fill out information (ID, date and time) on the sealed sticker attached to each can or inserted into the frozen pulses portion. In order to measure compliance, subjects will be asked to return all stickers at the end of the week, when new foods are provided to them. For those in the energy restriction group, the dietitian will a have a defined amount of time to advise on how to reduce caloric intake by 500 kcal per day at week 1 (the start of the study) and week 4 (halfway through the study). In addition, the dietitian will obtain a food history and ask additional pulse consumption questions at week 1 and week 8. Also, a 24 h food recall will be obtained from subjects by a dietitian at weeks 1, 4 and 8.

For all subjects, body weight, waist girth, blood pressure, fasting blood lipids, glucose, insulin and satiety hormones will be measured at weeks 1, 4 and 8. Each subject will arrive at the same chosen time for each session, between 8:00 and 10:00 a.m. Upon arrival, subjects will fill out a Sleep Habits and Stress Factors Questionnaire and a Food Intake and Activity Questionnaire. For each session, subjects will be asked to arrive after an overnight fast; only water will be allowed until 1 hour before blood collection.

Blood glucose and insulin response to a glucose load (75 g) will be determined at weeks 1 and 8. For this test (an oral glucose tolerance test), an indwelling catheter will be inserted in the antecubital vein by a nurse and blood samples will be taken at prior to (-15 minutes) and at 0, 10, 20, 30, 60, 90 and 120 minutes after the consumption of a 75 g glucose drink. A total of 90 ml of blood will be sampled at weeks 1 and 8. A single fasting blood sample (20 ml of blood) will also be obtained at week 4 for the same analysis. The week 1 and week 8 sessions will last a maximum of 4 hours and the week 4 session will last a maximum of 2 hours.

Blood samples will be analyzed for glucose, insulin, leptin, ghrelin, glucagon-like peptide-1 (GLP-1), low-density lipoprotein (LDL), triglyceride (TG), C-reactive protein, C-peptide, adiponectin and glycosylated hemoglobin (HbA1c).

Pulses will be obtained from Can Grow Foods, Heinz or purchased from the supermarket.

ELIGIBILITY:
Inclusion Criteria:

* overweight/obese adults
* body mass index: 27-35 kg/m2
* individuals not prescribed medications over the past 6 months that could interfere with the study outcomes (i.e. statins or metformin)

Exclusion Criteria:

* smokers
* those on an energy restricted diet
* breakfast skippers
* pregnant/lactating women

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
blood glucose, lipids and satiety hormones | 4 months

SECONDARY OUTCOMES:
body weight, waist circumference and blood pressure | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harvey G. Anderson, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- Leadership Sinai Centre for Diabetes, Mt. Sinai Hospital, Toronto, Ontario, Canada